CLINICAL TRIAL: NCT00838695
Title: Variability in Adrenergic Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, C. Michael Stein, Dan May Professor of Medicine, Professor of Pharmacology, Assistant Director of the Division of Clinical Pharmacology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 71148; P01HL056693 (NIH); 1UL1RR024975 (NIH)
Record Dates: First submitted 2009-02-04; First posted 2009-02-06 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Vascular Reaction to Medications
Keywords: Hand vein sensitivity; phenylephrine; nitroglycerin
MeSH Terms: interventions — Phenylephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- African Americans (Experimental): Subjects' hand veins will be measured for maximum constriction while being infused with phenylephrine, and then mental stress and cold pressor testing
  Interventions: Drug: Phenylephrine
- Caucasians (Experimental): Subjects' hand veins will be measured for maximum constriction while being infused with phenylephrine, and then mental stress and cold pressor testing
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Phenylephrine — Intravenous phenylephrine at low doses (approximately 10 doses ranging from 0-5000 ng/min) Intravenous nitroglycerin at low doses (approximately 10 doses ranging from 0.05-100 ng/min)
  Other Names: generic medications used,not applicable

SUMMARY:
The goal of this project is to determine the genetic factors contributing to interindividual differences in response to physiological and pharmacological vasoconstrictors and vasodilators.

DETAILED DESCRIPTION:
The dorsal hand vein model is a relatively non-invasive and robust experimental model to examine the local in vivo effect of vasoactive drugs without elucidating systemic counterregulatory reflexes. Infusion of incremental low doses of phenylephrine into a dorsal hand vein results in increasing local venoconstriction, without systemic effects. Similarly, infusion of incremental low doses of nitroglycerin into a preconstricted dorsal hand vein results in increasing local venodilation, without systemic effects. Systemic vascular responses can be measured by the cold pressor test (CPT),that leads to increase in blood pressure and heart rate , or mental stress that is also known to stimulate cardiovascular responses. Individuals vary in their local and systemic vascular responses but the genetic determinants of these are not clear.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years, inclusive.
* Subject must be willing to give written informed consent and be able to adhere to diet and study schedules.
* Subjects must be free of any clinically significant disease that requires a physician's care and/or would interfere with the study evaluations.
* Subjects must have a normal or clinically acceptable physical examination and ECG.
* Clinical laboratory tests (CBC, blood chemistries, and urinalysis) must be within normal limits or clinically acceptable to the investigator.

Exclusion Criteria:

* Any subject who has taken any prescription or over-the-counter drugs, other than oral contraception if female, within two weeks prior to study drug administration.
* Subjects who are presently, or were formerly, narcotic addicts or alcoholics.
* Subjects who have a clinically significant allergy/intolerance to phenylephrine.
* Females with a positive serum/urine pregnancy test at screening.
* Females who are nursing.
* Subject using sildenafil or other phosphodiesterase inhibitors.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles M Stein, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Result] Adefurin A, Ghimire LV, Kohli U, Muszkat M, Sofowora GG, Paranjape SY, Stein CM, Kurnik D. Blacks have a greater sensitivity to alpha1-adrenoceptor-mediated venoconstriction compared with whites. Hypertension. 2013 Apr;61(4):915-20. doi: 10.1161/HYPERTENSIONAHA.111.00854. Epub 2013 Feb 11. PMID 23399717
- [Result] Adefurin A, Ghimire LV, Kohli U, Muszkat M, Sofowora GG, Li C, Paranjape SY, Stein CM, Kurnik D. Genetic variation in the alpha1A-adrenergic receptor and phenylephrine-mediated venoconstriction. Pharmacogenomics J. 2015 Aug;15(4):310-5. doi: 10.1038/tpj.2014.69. Epub 2014 Nov 25. PMID 25421140
- [Result] Adefurin A, Ghimire LV, Kohli U, Muszkat M, Sofowora GG, Li C, Levinson RT, Paranjape SY, Stein CM, Kurnik D. Genetic variation in the alpha1B-adrenergic receptor and vascular response. Pharmacogenomics J. 2017 Jul;17(4):366-371. doi: 10.1038/tpj.2016.29. Epub 2016 Apr 19. PMID 27089938

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by advertisement within the Vanderbilt University campus and through the Vanderbilt University Clinical Research Center study volunteer database,
Period: Overall Study
Arm/Group | African Americans | Caucasians
Started | 42 | 64
Completed | 42 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | African Americans | Caucasians | Total
Number analyzed (Participants) | 42 | 64 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (8) | 26.9 (6.8) | 27 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 31 | 49
  Male | 24 | 33 | 57
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 64 | 106
plasma norepinephrine [Mean (Standard Deviation); unit: pg/ml] | 179.5 (70.8) | 162.3 (58) | 168.9 (63.2)
plasma epinephrine [Mean (Standard Deviation); unit: pg/ml] | 21.0 (15.6) | 18.5 (12.5) | 19.4 (13.7)

OUTCOME MEASURES:

1. Primary Outcome: ED50 After Phenylephrine
Description: ED50 is a measurement of vein constriction and indicates 50% of maximal constriction after being given medication phenylephrine, representing sensitivity to the drug. Phenylephrine was infused at increasing dose rates, ranging from 12-9600 ng/min. The infusion at each dose rate lasted 7 minutes, with the vein diameter measured during the last 2 minutes of the infusion. The number represents the ng/ml of phenylephrine needed to reach 50% of maximal vein constriction. ED50 values were not normally distributed and were log-transformed for analysis and expressed as geometric means.
Time Frame: 70 minutes
Measure: Geometric Mean (95% Confidence Interval); unit: ng/min
Arm/Group | African Americans | Caucasians
Number analyzed (Participants) | 42 | 64
ng/min | 172 [115 to 256] | 310 [222 to 434]

2. Secondary Outcome: Change in Blood Pressure
Description: change in systolic and diastolic blood pressure, comparing before and after cold pressor test. A subset of 57 participants (of the 106) who were in the primary outcome measure also participated in the cold pressor test.
Time Frame: baseline to 2 minutes
Population: A subset of participants (57 of the 106) in the primary outcome measure also participated in the cold pressor test.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | African Americans | Caucasians
Number analyzed (Participants) | 21 | 36
mmHg
  Change in Systolic Blood Pressure | 23.0 (12.3) | 18.9 (11.7)
  Change in Diastolic Blood pressure | 16.9 (9.3) | 16.4 (8.8)

ADVERSE EVENTS:
Time Frame: Adverse events were documented for participants from time they began diet of at least 4 days to end of study day.
Groups:
- African Americans: Participants who were of African American descent.
- Caucasians: Participants who were of Caucasian descent.
Arm/Group | African Americans | Caucasians
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/64
Other Adverse Events (participants affected / at risk) | 0/42 | 0/64

LIMITATIONS AND CAVEATS:
Findings derived from dorsal hand veins and cannot automatically be extrapolated to other vascular beds.

Women were not studied at predefined periods of menstrual cycle or account for use of hormonal contraceptives.

Some genotype groups were small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No